CLINICAL TRIAL: NCT06277869
Title: Testing the Role of Thermal Jacket in Attaining and Maintaining Euthermia Among Preterm and LBW Neonates in Clinical Setting of Bangladesh
Brief Title: Effectiveness Trial of Thermal Jacket
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other); Directorate General of Health Services (DGHS), Bangladesh (Unknown); Poeticgem International Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PR-22146
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Preterm Neonate; Low Birthweight Neonate
Keywords: Preterm neonate; Low birthweight neonate; Kangaroo Mother Care; Thermal Jacket
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal Jacket (Experimental): As a intervention, the enrolled preterm or low birthweight neonates gets the thermal jacket as well as Kangaroo Mother Care for thermal care.
  Interventions: Device: Thermal Jacket; Procedure: Kangaroo Mother Care
- Kangaroo Mother Care (Active Comparator): As a control, the enrolled preterm or low birthweight neonates gets the conventional Kangaroo Mother Care only.
  Interventions: Procedure: Kangaroo Mother Care

INTERVENTIONS:
Device: Thermal Jacket — In the intervention group, the enrolled preterm or low birthweight eligible neonates gets the intervention Thermal Jacket as well as Kangaroo Mother Care.
  Arms: Thermal Jacket
Procedure: Kangaroo Mother Care — Skin-to-Skin care, provided by primary caregiver.

SUMMARY:
Globally, over 15 million neonates are born preterm each year. They account for approximately 30% of global neonatal deaths and 19% of total neonatal deaths in Bangladesh. They usually die because they cannot maintain normal temperature due to their weight, immature skin and underdeveloped thermal regulatory capacity of the brain.

Maintaining continuous Kangaroo Mother Care (KMC) for at least 16-20 hours/day, is sometimes not feasible for mothers or caregivers. In addition, we also have the challenge of keeping preterm or low birthweight (LBW) neonates warm during transportation.

The scientists at icddr,b, Johns Hopkins University, and George Mason University developed the thermal jacket for keeping preterm or LBW neonate warm. We have already completed the laboratory trial on mannquins and clinical safety trial among preterm or LBW neonates. Now, we propose to build on our previous work by systematically testing the effectiveness trial of the 'thermal jacket' among preterm or LBW neonates at clinical settings.

Hypothesis: Thermal jacket can increase the rate of euthermia among the preterm or LBW neonates in the selected health facilities in Bangladesh.

Objectives: The aim of this study is to test whether the thermal jacket can attain and maintain euthermia of preterm or LBW neonates in clinical settings of Bangladesh.

DETAILED DESCRIPTION:
We will equip a cluster-randomized stepped-wedge trial design. We will select and onboard hospitals randomly from three districts in pre-intervention period which eventually go into post-intervention period. The study will be conducted in three phases. The pre-intervention period for eight weeks for baseline data collection. Then intervention period (introduce thermal jackets) for another 24 weeks, and post-intervention period for endline data collection for eight weeks. In the control phase, all the eligible neonates enrolled in the hospitals whose parents agree to participate in the study will be observed and monitored for their thermal status (euthermia, hypothermia, and hyperthermia). Once the hospitals shift to case phase the eligible neonates will be given with thermal jacket. The icddr,b team will observe and monitor the enrolled neonates' thermal status throughout the event period. For this study, the definition of an event is the data from an individual enrolled infant on six hours' basis. Thus, every twenty-four hours, we can collect four events from a single neonate. During thermal care uptake, let it be with KMC or thermal jacket, the axillary temperature of the enrolled neonates will be recorded every 60 minutes. Feeding history will be recorded until discharge. According to the national newborn health SOP, during both control and case phases, mothers will be encouraged to provide KMC. The thermal jacket will be offered to mother when KMC will be ceased or not given by the neonate's family members. The thermal jacket intervention will be ceased for each neonate if mother wants to provide KMC or doesn't wish to put the neonate on the thermal jacket anymore. Thermal jacket will be provided for the time period as long as mother or legal guardian wishes to keep their neonate in the jacket without any time limitation. Mothers or caregivers of each neonate will be provided with training on KMC and thermal jacket and due support during the uptake of the KMC and thermal jacket will be provided as well. The data those will be collected during the pre-phase will be the control data and data that will be collected during the post-phase will be the intervention data.

ELIGIBILITY:
Inclusion Criteria:

1. KMC eligible neonates
2. Heart rate 100-160 per minute
3. Capillary Refill Time ≤ 3 sec
4. Respiratory rate 30-59 per minute
5. Breaths comfortable
6. Pink in room air

Exclusion Criteria:

1. In nasogastric tube
2. In oxygen therapy
3. In intravenous fluid
4. Sign of respiratory distress
5. Prolonged or frequent apnea
6. Major surgical problem
7. Gross congenital anomaly

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Body temperature of preterm or low birthweight neonates maintain the euthermic range. | 6 hours per event
  The primary outcome of this phase is attainment and maintenance of euthermia, defined as i. Having reached to 36.5⁰ C for hypothermic neonates at any point of a single event, ii. Maintaining euthermia throughout the event and iii. Having risen the temperature up to the euthermic range within 1 hour if at any point neonate goes below euthermic range. The endpoint of each event will be ascertained for every neonate during the pre-phase and intervention-phase in the same manner regardless of whether the thermal jacket is used.

CONTACTS AND LOCATIONS:
Overall Officials: Anisuddin Ahmed, MS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (3):
- Bangladesh (3):
  - Lakshmipur District Hospital, Lakshmīpur, Chattogram
  - Kushtia 250 Bedded General Hospital, Kushtia, Khulna Division
  - Jamalpur 250 Beded General Hospital, Jamālpur, Mymensingh